CLINICAL TRIAL: NCT03795467
Title: Association Between the Peripheral Perfusion Index, Haemoglobin Levels and Blood Transfusions in Patients Undergoing Acute Abdominal- and Orthopaedic Surgery.
Brief Title: Peripheral Perfusion Index, Haemoglobin and Blood Transfusion in Acute Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Agerskov, MD, Research Fellow, Hvidovre University Hospital
Record Dates: First submitted 2019-01-02; First posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Fracture of Hip; Ileus; Perforated Viscus; Anastomotic Leak
MeSH Terms: conditions — Hip Fractures; Ileus; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The peripheral perfusion index (PPI) is a non-invasive, feasible measure of peripheral perfusion and, assumed, the overall circulation, which all patients are monitored by.

This study is carried out to assess the association between values of PPI, haemoglobin and blood transfusion.

Hypothetically, patients with low values of hb are more susceptible to a deteriorating circulation reflected in poorer PPI regardless of blood pressure and that resuscitation with blood products improves PPI measurements. Moreover, that patients with low values of PPI have more surgical complications and higher mortality.

DETAILED DESCRIPTION:
Background: Acute surgical patients with e.g. hip fracture (HF) or acute abdominal surgical conditions often have comorbidities and a fragile circulation. Haemodynamic challenges make these patients vulnerable during anaesthesia, and perioperative complications are frequent.

Anaemia is associated with increased mortality and adverse outcomes in patients undergoing surgery. One of the consequences of acute anaemia is reduced blood oxygen content, leading to reduced tissue oxygen delivery and development of tissue hypoxia. Patients with e.g. HF have a large drop in haemoglobin (hb) level that occurs after the injury, yet prior to the surgery. It is therefore important to be aware of the risk of preoperative anaemia even when the initial hb levels appear to be normal. Perioperative hb are associated with shorter lengths of hospital stay, reduced mortality and lower readmission rates, and patients with postoperative anaemia have increased mortality and length of hospital stay.

Haemodynamic monitoring is traditionally based on measurement of blood pressure (BP) and heart rate (HR) but these measurements may be insufficient in evaluating overall oxygen delivery and perfusion of vital organs. An apparently sufficient BP and, for patients with more specialised monitoring, cardiac output (CO), does not necessarily mean a sufficient peripheral microcirculatory flow due to compensatory mechanisms, but on the other hand a low CO may be sufficient in context of low metabolic demand.

The non-invasive peripheral perfusion index (PPI) is a numerical value of peripheral perfusion measured by the pulse oximeter derived from the photoelectric plethysmographic signal. PPI is represents the ratio between the pulsatile component (arterial) and the non-pulsatile component (venous blood, capillary blood and other tissues) of the light reaching the detector of the pulse oximeter, and reflects changes in peripheral blood flow as the pulsatile component increases with vasodilatation and decreases with vasoconstriction. It is an accessible way to obtain a measure for peripheral perfusion as pulse oximeters are universally available in all operating rooms and intensive care units. Previous studies have shown that PPI is a useful indicator of reduced peripheral blood flow both in clinical and experimental settings. Correlation between clinical symptoms of reduced peripheral perfusion such as low temperature, increased capillary response and reduced PPI in critically ill patients has been demonstrated, and a reduced peripheral perfusion may be a predictor of mortality and complications in patients undergoing major surgical procedures and in septic shock patients.

Hypothetically, patients with low values of hb are more susceptible to a deteriorating circulation reflected in poorer PPI regardless of blood pressure and that resuscitation with blood products improves PPI measurements. Moreover, that patients with low values of PPI have more surgical complications and higher mortality.

Method: The main objective of this study is to estimate the association between perioperative values of PPI and haemoglobin levels. The secondary objectives are to evaluate PPI in patients with low hb in relation to mean arterial blood pressure (MAP), and evaluate changes in PPI with patients with low and normal hb in relation to transfusion with blood products.

ELIGIBILITY:
Inclusion Criteria:

* Orthopedic surgery patients with fracture of the hip, booked in the electronic patient record for operation with procedural codes:KNFB02 HNFJ81 KNFJ51 KNFJ52 KNFJ70
* Acute abdominal surgery patients booked in the electronic patient record for operation with procedural codes:KJAH01 KJAH00

Exclusion Criteria:

* No sampling of PPI registered
* Foreign/temporary civil registration number
* Already included in cohort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 18 years of age having performed acute abdominal or orthopedic surgery from 1th November 2017 through 31th October 2018 at Hvidovre and Bispebjerg University Hospitals. Study subjects will be obtained from the hospitals electronic medical records via specific procedural- or diagnostic codes representing the acute orthopedic or abdominal surgery in the specified one-year period.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Peripheral perfusion index | Perioperative with 5 minute interval
  Absolute PPI levels
Haemoglobin level | Time interval: From 3 hours preoperative to 10 hours postoperative
  Measurement of haemoglobin by blood sample or artery gas.

SECONDARY OUTCOMES:
Evaluation of Peripheral perfusion index in patients with high vs. low haemoglobin levels in relation to mean arterial blood pressure (MAP). | Perioperative
  High vs. low hb defined as 6,0 < hb > 6,0. Absolute PPI levels perioperative with a 5 minute interval. Absolute values of MAP measured perioperative with a 5 minute interval.
Proportion of transfusion with blood products in patients with perioperative high vs. low haemoglobin levels. | Perioperative
  High vs. low hb defined as 6,0 < hb > 6,0. Blood transfusion measured as total amount used perioperatively.
Evaluation of peripheral perfusion index changes in patients with perioperative high vs. low haemoglobin levels in relation to transfusion with blood products . | Perioperative
  High vs. low hb defined as 6,0 < hb > 6,0. Absolute PPI levels perioperative measured with a 5 minute interval. Blood transfusion measured as total amount used perioperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia, Hvidovre Hospital, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lau FF, Agerskov M, Thusholdt ANW, Hojlund J, Meyhoff CS, Jans O, Foss NB. Peripheral perfusion index stratifies risk in patients with intraoperative anemia: A multicentre cohort study. J Clin Anesth. 2024 Aug;95:111472. doi: 10.1016/j.jclinane.2024.111472. Epub 2024 Apr 12. PMID 38613938